CLINICAL TRIAL: NCT07185516
Title: Airway Ultrasound Indices Versus Clinical Assessment for Prediction of Difficult Laryngoscopy in Elective Surgical Pediatric Patients
Brief Title: Airway Ultrasound Indices for Prediction of Difficult Laryngoscopy in Pediatric Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, assistant professor, Ain Shams University
Other Study IDs: FMASU MD57/2023
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Airway Ultrasound Indices; Clinical Airway Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway assessment: clinical and ultrasound assessment of the airway
  Interventions: Other: Airway ultrasound indices; Other: Clinical airway assessment

INTERVENTIONS:
Other: Airway ultrasound indices — Tongue thickness, hyomental distance in neutral position (HMDRn), hyomental distance in extended position (HMDRe), ratio of hyomental distance in both positions (HMDR), thyromental distance (TMD), ratio of tongue thickness to thyromental distance (TT/TMD), epiglottis thickness &pre-epiglottic space thickness
Other: Clinical airway assessment — Mallampati grading and thyromental distance (TMD). The glottic structures displayed during laryngoscopy will be classified according to the Cormack-Lehane

SUMMARY:
The goal of this observational study is to compare the airway ultrasound indices and the preoperative clinical airway assessment concerning the difficult laryngoscopic view in paediatric patients undergoing elective surgery under general anaesthesia

The main question it aims to answer is:

• Do airway ultrasound indices better predict difficult laryngoscopic view in paediatric patients than clinical airway assessment?

DETAILED DESCRIPTION:
Airway-related morbidity, as a result of an inability to anticipate a difficult airway, remains the primary concern for an anesthesiologist. Various clinical measurements and methods, such as the thyromental distance (TMD), sternomental distance, horizontal length of the mandible, head and neck movement, and the Mallampati score, were used to predict difficult laryngoscopy and intubation in adult patients. However, using these measurements in the pediatric population is not as easy as in adults.

The use of airway sonography has been extended as an assessment tool for a difficult airway. Various parameters like tongue thickness, anterior soft tissue thickness, and hyomental distance ratio have been used to predict a difficult airway. However, the usefulness of ultrasonography to predict a difficult airway in infants and children has still not been described. This study will compare the effectiveness of clinical measurements to the ultrasound indices in predicting difficult laryngoscopic view in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I and II.
* Patients undergoing elective surgery under general anaesthesia

Exclusion Criteria:

* Congenital upper airway malformation.
* Head and neck swellings.
* Scars.
* Radiation to the neck.
* Tracheotomy.
* Neurosurgical or cardiac procedures.
* ENT surgeries.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric patients aged 7 to 12 years old of both sexes undergoing elective surgery under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of difficult intubation | 60 Seconds
  failure to intubate the patient within 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Hussien, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided